CLINICAL TRIAL: NCT03644602
Title: Beneficial Effects of a Low FODMAPs Diet in Different Gastrointestinal Disorders
Brief Title: Low FODMAPs Diet in Gastrointestinal Disorders
Acronym: FODMAPs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Fabiana Castiglione, Associate Professor, Federico II University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 285/16
Record Dates: First submitted 2017-07-04; First posted 2018-08-23 (Actual); Last update posted 2018-08-23 (Actual); Status verified 2018-08

CONDITIONS: Inflammatory Bowel Diseases; Irritable Bowel Syndrome; Coeliac Disease
Keywords: low FODMAPs diet; Adherence; Inflammatory Bowel Diseases; Irritable Bowel Syndrome; Coeliac Disease
MeSH Terms: conditions — Inflammatory Bowel Diseases; Irritable Bowel Syndrome; Celiac Disease | interventions — FODMAP Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- IBD patients (Active Comparator): All subjects with Crohn's disease in clinical remission (defined in the presence of a Crohn's Disease Activity Index, CDAI <150), and with Ulcerative colitis in clinical remission (defined in the presence of <3 evacuations / day without blood, in the absence of endoscopic alterations) received a low FODMAPs diet.
  The low FODMAPs diet was administered for 3 months.
  Interventions: Dietary Supplement: low FODMAPs diet
- Coeliac patients (Active Comparator): Celiac patients on a gluten free diet for at least one year received a low FODMAPs diet. The low FODMAPs diet was administered for 3 months.
  Interventions: Dietary Supplement: low FODMAPs diet
- IBS patients (Active Comparator): Patients with Irritable Bowel Syndrome received a low FODMAPs diet. The low FODMAPs diet was administered for 3 months.
  Interventions: Dietary Supplement: low FODMAPs diet

INTERVENTIONS:
Dietary Supplement: low FODMAPs diet — Low FODMAPs diet was a diet containing low amount of poorly absorbed short-chain carbohydrates (Fermentable, Oligo-, Di-, Mono-saccharides And Polyols)

SUMMARY:
Recent studies have shown that FODMAPs (Fermentable Oligosaccharides, Disaccharides, Monosaccharides, and Polyols) free diet is efficient in subjects with Irritable Bowel Syndrome (IBS). Patients with Inflammatory Bowel Diseases (IBD) and celiac disease (CD) can experience functional gastrointestinal symptoms not related to inflammation, but data about the use of low FODMAPs diet in these settings are still scarce. The aim of the present study was to evaluate the usefulness of a low FODMAPs diet in patients with IBS, non-active IBD and CD on strict gluten-free diet (GFD). A low FODMAPs diet could be a valid option to contrast abdominal symptoms in patients with IBS, non-active IBD and CD on GFD, thus improving the quality of life and the social relations.

DETAILED DESCRIPTION:
Recurrent gastrointestinal symptoms (bloating, constipation, abdominal pain, diarrhea and flatulence) often interfere with patients' quality of life (QoL) and daily activities. These symptoms have been noted in various diseases such as irritable bowel syndrome (IBS), celiac disease (CD) and inflammatory bowel diseases (IBD). IBS is the most common diagnosis made by gastroenterologists and affects up to 15% of the population. About 60% of patients with IBS claims that certain foods can exacerbate their symptoms, so pharmacological treatment is often accompanied by dietary measures. Very recently, a diet for the management of functional symptoms associated with IBS has been developed: the low FODMAPs diet. FODMAPs (Fermentable, Oligo-, Di-, Mono-saccharides And Polyols) is a collective term that indicates a family of poorly absorbed short-chain carbohydrates. The low FODMAPs diet is a relatively novel area of interest and the majority of studies have been performed in patients with IBS; most of them showed that limiting FODMAPs led to an improvement of intestinal symptoms. Patients with Crohn's disease (CrD) and ulcerative colitis (UC) often experience symptoms related to concomitant functional disease, such as bloating, abdominal pain and flatulence, in the absence of active inflammation. These symptoms are less likely to respond to the common anti-inflammatory drugs and it is important to recognize them, in order to avoid inappropriate therapy and improve QoL. In effect, the cause of these symptoms is related to altered function of the gut and the enteric nervous system, rather than to the inflammatory activity of disease. In these patients, carbohydrate malabsorption has been considered a candidate mechanism by which the diet can induce gut symptoms: lactose and fructose malabsorption has been recognized as a potential cause of symptoms due to the high osmotic activity and fermentability of malabsorbed lactose.

The management of this condition could benefit of a dietary intervention, but data regarding the effect of a low FODMAPs diet in IBD are limited.

Also in coeliac patients, despite a lifelong GFD, some abdominal symptoms such as flatulence, bloating, diarrhea and abdominal pain can persist. However data regarding the effect of a low FODMAPs diet in these subjects are still scarce.

On the basis of these considerations, the aim of this study was to evaluate the clinical impact of a low FODMAPs diet in patients with IBS, CD on GFD and IBD in remission.

Each subject who respected the inclusion criteria was enrolled in the study and was submitted to a diet low in FODMAPs content, after filling out questionnaires on quality of life and symptoms (IBS-SSS and SF-36) (T0).

The IBS-SSS questionnaire consists of 5 questions on: the severity and frequency of abdominal pain, the severity of the bloating, the level of satisfaction in bowel habits and quality of life. Patients give an estimate from 0 to 100 and the results of each question are summed to obtain the final score (theoretical range of 0-500, with a higher score indicating worse condition). Previous studies have established that scores below 175 represents mild IBS symptoms, 175-300 represents moderate severity, and scores above 300 represent severe IBS.

The SF-36 is a questionnaire on the patient's state of health consisting of 36 questions related to eight health domains: AF-physical activity (10 questions), RP-role limitations due to physical health (4 questions) and RE-role limitations due to emotional problems (3 questions), BP-physical pain (2 questions), GH-perception of general health (5 questions), VT-vitality (4 questions), SF-social activities (2 questions), MH-mental health (5 questions) and a single question about the change in health status. All SF-36 questions, except one, are referred to a previous four-week period of the compilation of questionnaire. The eight-scaled scores are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight: the lower the score the more disability; the higher the score the less disability.

After the administration of the questionnaires and the collection of anthropometric measurements (weight and height), patients were put on a low FODMAPs diet (T0). Each regimen was specific for the patient's energy requirement (calculated by BMI) and for its content in FODMAPs, realized in conformity with the food reference tables. This low FODMAPs diet was prescribed by a dietitian for 12 weeks and patients were instructed to eat according to their appetite, received a summary diagram with substances to be taken and those to be avoided and were educated to interpret food labels/ingredients lists.

In order to cover the needs of micro and macronutrients, the administered dietary patterns maintained the contents of oligosaccharides, fructose and polyols not more than 0.5 g.

The questionnaires and the clinical evaluation of the patients were repeated one month (T1) and three months (T3) after the beginning of the diet.

ELIGIBILITY:
Inclusion Criteria:

* IBS patients
* IBD patients in remission
* Coeliac patients on gluten free diet

Exclusion Criteria:

* Active IBD
* Coeliac patients non compliant to gluten free diet

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Improvement of IBS-SSS after 3 months | 1 month and 3 months
  to evaluate the clinical impact of a low FODMAPs diet in patients with IBS, CD on GFD and IBD in remission. Each subject who respected the inclusion criteria was enrolled in the study and was submitted to a diet low in FODMAPs content, after filling out questionnaire on quality of life and symptoms (IBS-SSS).
  The questionnaire was re-administered after 1 month and 3 months of low FODMAPs diet.

SECONDARY OUTCOMES:
Improvement of SF-36 after 3 months | 1 month and 3 months
  to evaluate the clinical impact of a low FODMAPs diet in patients with IBS, CD on GFD and IBD in remission. Each subject who respected the inclusion criteria was enrolled in the study and was submitted to a diet low in FODMAPs content, after filling out questionnaire on quality of life and symptoms (SF-36).
  The questionnaire was re-administered after 1 month and 3 months of low FODMAPs diet.

CONTACTS AND LOCATIONS:
Overall Officials: Fabiana Castiglione, Principal Investigator — Federico II University
Locations (1):
- Aou Federico Ii, Naples, Italy

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-07-20): https://cdn.clinicaltrials.gov/large-docs/02/NCT03644602/Prot_SAP_000.pdf
  • Informed Consent Form (2017-07-20): https://cdn.clinicaltrials.gov/large-docs/02/NCT03644602/ICF_001.pdf